CLINICAL TRIAL: NCT03609255
Title: Health Effects of Reducing Sedentary Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Martin Binks, Associate Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TTUIRB2018-347
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: General Population

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (C) (Active Comparator)
  Interventions: Behavioral: Control
- Sedentary behavior group (SB) (Experimental)
  Interventions: Behavioral: Reducing sedentary behavior
- Stress management group (SR) (Experimental)
  Interventions: Behavioral: Reducing stress

INTERVENTIONS:
Behavioral: Reducing sedentary behavior — Educational handouts for sedentary behavior and strategies reducing sedentary behavior and weekly videos related to reduced sedentary behavior
  Arms: Sedentary behavior group (SB)
Behavioral: Reducing stress — Educational handouts for sedentary behavior and stress management handout and weekly videos related stress management
  Arms: Stress management group (SR)
Behavioral: Control — An educational handout for sedentary behavior and weekly neutral topic videos
  Arms: Control group (C)

SUMMARY:
A recent review indicated that sedentary behavior has been associated with increased morbidity and mortality but the intervention studies frequently focus only on changing sedentary behavior (reducing sedentary time) without measuring health-associated outcomes. Elevated cortisol (related to stress) has been linked with health risks. Improved physical fitness has been linked with improved cortisol responses to psychosocial stressors. In addition, increased physical activity induced favorable effects upon low density lipoprotein, high density lipoprotein, and total cholesterol. Previous study also indicated that increasing daily steps have positive effect on blood glucose in people with impaired glucose tolerance. Ultimately, the investigators think that sedentary intervention and stress management may have benefits on these health indicators. As such the investigators will examine whether sedentary intervention or stress management can have positive effect on human health by measuring salivary cortisol, blood lipid profile, fasting blood glucose, blood pressure, resting energy expenditure, and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years.

Exclusion Criteria:

* Unable/unwilling to provide informed consent.
* Having mobility impairment.
* Current severe untreated depression (i.e., score in the severe depression range on the Hospital Anxiety and Depression Scale; HADS).
* Women who are pregnant or nursing.
* Currently smoking (within last 12 months).
* Currently use medications that affect salivary cortisol level (i.e. prednisone, dexamethasone).
* Have been diagnosed Addison's disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Daily steps | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in daily steps measured via pedometer.
Stress improvement in sedentary behavior group (SB) | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Improvement in stress as measured via Perceived Stress Scale (PSS) in SB.
Stress improvement in sedentary behavior group (SB) | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Improvement in stress as measured via salivary cortisol in SB.
Stress improvement in stress management group (SR) | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Improvement in stress as measured via Perceived Stress Scale (PSS) in SR.
Stress improvement in stress management group (SR) | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Improvement in stress as measured via salivary cortisol in SR.
Compare the changes of stress levels between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compare the changes of stress levels as measured via Perceived Stress Scale (PSS) between SB and SR.
Compare the changes of stress levels between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compare the changes of stress levels as measured via salivary cortisol between SB and SR.

SECONDARY OUTCOMES:
Changes in low density lipoprotein (LDL) in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in LDL as measured via finger stick in SB.
Changes in high density lipoprotein (HDL) in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in HDL as measured via finger stick in SB.
Changes in total cholesterol (TC) in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in TC as measured via finger stick in SB.
Changes in triglyceride (TG) in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in TG as measured via finger stick in SB.
Changes in fasting blood glucose in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in fasting blood glucose as measured via finger stick in SB.
Changes in body fat in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in body fat as measured via BODPOD in SB.
Changes in weight in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in weight as measured via BODPOD in SB.
Changes in blood pressure in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in blood pressure as measured via Omron Digital BP Monitor HEM-907XL in SB.
Changes in low density lipoprotein (LDL) in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in LDL as measured via finger stick in SR.
Changes in high density lipoprotein (HDL) in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in HDL as measured via finger stick in SR.
Changes in total cholesterol (TC) in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in TC as measured via finger stick in SR.
Changes in triglyceride (TG) in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in TG as measured via finger stick in SR.
Changes in fasting blood glucose in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in fasting blood glucose as measured via finger stick in SR.
Changes in body fat in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in body fat as measured via BODPOD in SR.
Changes in weight in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in weight as measured via BODPOD in SR.
Changes in blood pressure in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Changes in blood pressure as measured via Omron Digital BP Monitor HEM-907XL in SR.
Compared the changes in LDL between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compared the changes in LDL between SB and SR.
Compared the changes in HDL between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compared the changes in HDL between SB and SR.
Compared the changes in TC between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compared the changes in TC between SB and SR.
Compared the changes in TG between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compared the changes in TG between SB and SR.
Compared the changes in fasting blood glucose between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compared the changes in fasting blood glucose between SB and SR.
Compared the changes in body fat between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compared the changes in body fat between SB and SR.
Compared the changes in weight between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compared the changes in weight between SB and SR.
Compared the changes in blood pressure between SB and SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Compared the changes in blood pressure between SB and SR.
Change in resting energy expenditure in SB | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Change in resting energy expenditure as measured by metabolic cart in SB.
Change in resting energy expenditure in SR | Baseline (pre-intervention) and 4 weeks (post-intervention)
  Change in resting energy expenditure as measured by metabolic cart in SR.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas, United States